CLINICAL TRIAL: NCT04813419
Title: Efficacy and Safety Comparison Between Fractional 2940nm Er:YAG Laser and Fractional 1927nm Thulium Laser in the Treatment of Facial Atrophic Acne Scars
Brief Title: 2940nm Er:YAG Laser and 1927nm Thulium Laser in Improving Atrophic Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0227
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Atrophic Acne Scar
Keywords: 2940nm Er:YAG laser, 1927nm thulium laser
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: adult patients with similar atrophic acne scar on both sides of face
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and outcomes assessor are blinded to laser therapy received at each side of face
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- right face (Active Comparator): The right side of face of subjects
  Interventions: Device: 2940nm Er:YAG laser
- left face (Experimental): The left side of face of subjects
  Interventions: Device: 1927nm thulium laser

INTERVENTIONS:
Device: 1927nm thulium laser — The right face of subjects were treated with fractional 2940nm Er:YAG laser(MCL 31 Asclepion Laser Technologies, Germany), N25 mode. Energy was adjusted from 12 to 27J according to the severity of scarring. The left face of subjects were treated with fractional 1927nm thulium laser(Lavieen, korea). Parameters were set as stamp mode, a spot size of 5*5mm, a pulse time of 1000us, an energy intensity of 3645mJ/cm2 and a repetition of 1-3 times. All patients received 3 treatment sessions totally at an average interval of 4 to 6 weeks.
  Arms: left face
Device: 2940nm Er:YAG laser — The right face of subjects were treated with fractional 2940nm Er:YAG laser(MCL 31 Asclepion Laser Technologies, Germany), N25 mode. Energy was adjusted from 12 to 27J according to the severity of scarring. All patients received 3 treatment sessions totally at an average interval of 4 to 6 weeks.
  Arms: right face

SUMMARY:
Fractional non-ablative laser (FNAL) has been widely used in improving acne scarring. However, there was only one study reported efficacy and safety of the fractional non-ablative 1927nm thulium laser (FTL) and no studies have reported a comparison between FTL and fractional ablative 2940nm Er:YAG laser(FEL), which had been proved effective and safety in many studies. Thus, we designed a prospective, simultaneous spilt-face trial to evaluate the efficacy and safety of FTL in the treatment of acne scarring and make a comparison between FTL and FEL, hoping to provide a new available modality for patients who are intolerable or reluctant to ablative lasers.

DETAILED DESCRIPTION:
Acne vulgaris is a chronic and recalcitrant inflammation of pilosebaceous unit that has a high incidence rate in adolescence and even adults. Acne scarring is not an uncommon cosmetic complication which will cause physical and phycological pressure and impair the life quality of patients. It can be divided into two types according to morphology: atrophic and hypertrophic acne scarring. Atrophic acne scarring can be subclassified into boxcar, icepick and rolling scarring due to morphological features. Although a great variety of modalities to treat atrophic acne scarring such as chemical peeling, lasers and light, micro-needling and radiofrequency have emerged, fractional laser (FL) have come out on top. Unlike resurfacing lasers, FL creates three-dimensional, evenly distributed "microscopic thermal zones(MTZs)"on the treating area, which only covering about 3-40% of the skin and leaving the surrounding tissue undamaged and serving as "cell reservoir". Then, the MTZs can be rapidly replaced by keratinocytes in "cell reservoir" within the first 24 hours and by new collagen within 3-6 months. FL can be categoried into fractional ablative laser(FAL) and fractional non-ablative laser(FNAL).

With a wavelength of 2940nm, FEL could be highly absorbed by water-containing tissues of skin and cause superficial epidermis ablation and collagen induction[4]. But thermal damage is limited to about 20-50um. FTL has a moderate affinity for water content tissue. Thus, rather than causing epidermis turnover, it keeps the epidermis intact. But it can penetrate deep into 200-300um and stimulate collagen regeneration. Prior studies have shown that both FAL and FNAL were effective in treating acne scarring and the former were more effective while the latter had less side effects. However, in our clinic, we have observed outstanding effect and high satisfaction rate of FTL in improving atrophic acne scarring. Since there was only one clinical trial reported the efficacy and safety of FTL in Asian and no study have made a comparison between FTL and FEL, we designed this prospective, simultaneous spilt-face trial, hoping to provide a new available modality for patients who are intolerable or reluctant to ablative lasers.

ELIGIBILITY:
Inclusion Criteria:

age of at least 18 years clinical diagnose of facial atrophic acne scarring

Exclusion Criteria:

there was infection in the treatment site Acne vulgaris were not controlled had a propensity for keloid forming received oral isotretinoin or laser treatment in the past 3 months received chemical peeling 1 month before the study pregnancy or breast-feeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Goodman＆Baron quantitative global scarring grading system (GBS) | GBS change from baseline(T0) at 1 hour before the third session(T1) and 3 months after the final treatment(T2)
  It is evaluated by a blinded dermatologist. It is a international criteria evaluating acne scar according to scar number and type. Tpye :(A) Milder scarring(1 point each): macular erythematous or pigmented and mildly atrophic dish-like;(B)Moderate scarring(2 points each) :moderately atrophic dish-like, punched out with shallow bases, small scarring(<5mm), shallow but broad atrophic areas;(C)Severe scarring(3 points each): punched out with deep but normal bases, small scarring(<5mm), punched out with deep abnormal bases, small scarring(<5mm), linear or troughed dermal scarring, deep, broad atrophic areas. Scar numbers:1-10(1 point each), 11-20(2 points each),>20(3 points each).
self-rated acne scar improvement | 3 months after the final treatment(T2)
  It is evaluated by subjects themselves. Self-rated acne scar improvement ranged from 0 to 4, 0 meant no improvement, 1 represented 1-25% improvement, 2 represented 26-50% improvement, 3 represented 51-75% improvement and 4 represented 76-100% improvement.
self-rated satisfaction score | 3 months after the final treatment(T2)
  It is evaluated by subjects themselves. Satisfaction score ranged from 0 to 10: 0 meant not satisfied and 10 meant very satisfied.

SECONDARY OUTCOMES:
Pain score | immediately after each laser treatment
  It is evaluated by subjects themselves with Visual analogue scale(VAS) , on a scale from 0 to 10, 0 meant no pain while 10 meant extremely painful.

OTHER OUTCOMES:
adverse effects | through study completion, an average of 0.5 year
  Adverse reactions such as pain, erythema and edema, hyperpigmentation and hypopigmentation were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suiqing S Cai, doctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Since the individual participant data(IPD) is personal information, our participants are unwilling to share. But we welcome any questions through emails.